CLINICAL TRIAL: NCT00509054
Title: Randomised Clinical Trial of the Use of a Prosthetic Mesh to Prevent Parastomal Hernia
Brief Title: Prevention of Parastomal Hernia With a Mesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sundsvall Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Preventing parastomal hernia
Record Dates: First submitted 2007-07-30; First posted 2007-07-31 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2001-01

CONDITIONS: Parastomal Hernia
Keywords: Parastomal hernia, wound infection, stoma care.
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Prophylactic mesh — A low weigth partly absorbable mesh in a subaly posistion
  Other Names: Vypro mesh, Ethicon.

SUMMARY:
Parastomal hernias are randomised to either a conventional stoma formed through the rectus anterior muscle or to the same procedure with the addition of a prophylactic mesh in a sublay position.

DETAILED DESCRIPTION:
Parastomal hernias are randomised to either a conventional stoma formed through the rectus anterior muscle or to the same procedure with the addition of a prophylactic mesh in a sublay position. Randomisation is by opening closed envelopes.

A low-weight,partly absorbable mesh is used. Patients are followed for 5 years. Clinical follow up after one month to register early complications such as wound infection or mesh infection.

Clinical follow up after 12 months to register parastomal herniation, fistula formation, stenosis.

Clinical follow up after 5 years to register parastomal herniation, fistula formation, stenosis. At this clinical follow up radiologic examination is added.

ELIGIBILITY:
Inclusion Criteria:

* Clinical need of an enterostoma

Exclusion Criteria:

* Patients denies inclusion in the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2001-01; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Wound infection,mesh infection, parastomal hernia. | Within five years

SECONDARY OUTCOMES:
Fistula formation, stenosis,pain. | Within five years

CONTACTS AND LOCATIONS:
Overall Officials: Leif A Israelsson, MD,PhD, Study Director — Umea University
Locations (1):
- Kirurgkliniken Sundsvalls sjukhus, Sundsvall, Sweden

REFERENCES:
- [Result] Janes A, Cengiz Y, Israelsson LA. Preventing parastomal hernia with a prosthetic mesh. Arch Surg. 2004 Dec;139(12):1356-8. doi: 10.1001/archsurg.139.12.1356. PMID 15613293